CLINICAL TRIAL: NCT03126799
Title: A Randomized Phase II Study of Erlotinib Alone Versus Erlotinib Plus Bevacizumab for Advanced Non-small Cell Lung Cancer With Epidermal Growth Factor Receptor Activating Mutations
Brief Title: A Study of Tarceva vs. Avastin+Tarceva for Advanced NSCLC With EGFR m(+)
Acronym: AvaTa
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Roche Korea co.,Ltd. (Unknown)
Responsible Party: Principal Investigator, Ji-youn Han, Head of Center for Lung Cancer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC-2016-0107
Record Dates: First submitted 2017-03-30; First posted 2017-04-24 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: EGFR Positive Non-small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Erlotinib only (Active Comparator): Standard therapy arm:
  Erlotinib 150mg. po, qd, daily, q 3weeks
  Interventions: Drug: Erlotinib
- B: Erlotinib plus Bevacizumab (Experimental): Study treatment arm; Erlotinib 150mg, po. qd, daily, q 3weeks plus Bevacizumab 15mg/kg, iv, on D1, q 3weeks.
  Interventions: Drug: Erlotinib plus Bevacizumab

INTERVENTIONS:
Drug: Erlotinib plus Bevacizumab — Erlotinib 150mg, po, daily, q 3weeks plus Bevacizumab 15mg/kg, IV, on D1 Q 3 weeks
  Other Names: Tarceva plus Avastin
  Arms: B: Erlotinib plus Bevacizumab
Drug: Erlotinib — Erlotinib 150mg, po, daily, Q weeks
  Other Names: Tarceva
  Arms: A: Erlotinib only

SUMMARY:
Korean data of treating EGFR mutation positive NSCLC patients with Erlotinib and Bevacizumab is significantly necessary for developing new standard treatment in first-line therapy in Korean EGFR mutant NSCLC patients.

In this study, The investigators will investigate the efficacy and safety of Erlotinib and Bevacizumab combination compare to Erlotinib alone in Korean EGFR-mutant NSCLC patients.

DETAILED DESCRIPTION:
EGFR-TKIs are the standard first-line treatment option for EGFR-mutant NSCLC. After a randomized phase II trial, JO25567 was presented at 2014 ASCO, the synergistic effect of progression-free survival(PFS) could be expected when EGFR TKI, Erlotinib is combined with Antiangiogenesis agent, Bevacizumab. Even Korean and Japanese are classified as Asian based on location, the figure of Korean is more tended to Western people due to the dietary life in recent years. However the incidence rate of EGFR mutation positive patients in Korea is much higher than Western countries.

Therefore Korean data of treating EGFR mutation positive NSCLC patients with Erlotinib and Bevacizumab is significantly necessary for developing new standard treatment in first-line therapy in Korean EGFR mutant NSCLC patients.

In this study, The investigators will investigate the efficacy and safety of Erlotinib and Bevacizumab combination compare to Erlotinib alone in Korean EGFR-mutant NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed stage IIIB & IV non-small cell lung cancer other than squamous cell carcinoma
* Patients with one or more measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
* Locally diagnosed sensitive EGFR mutation positive (Exon 19 deletion or L858R)
* ECOG performance 0~1
* Age ≥ 19 years and - No previous treatment

Adequate organ function by following:

* ANC ≥1,500/uL, hemoglobin ≥9.0g/dL, platelet ≥100,000/uL
* Serum bilirubin < 1 x UNL, AST (SGOT) and ALT (SGPT) < 2.5 x UNL, If Liver metastasis, Serum bilirubin < 3 x UNL, AST (SGOT) and ALT (SGPT) < 5 x UNL
* Serum Cr ≤ 1 x UNL
* Patients who have had undergone radiotherapy are acceptable if patients meet all of the following criteria:

  * No history of irradiation to pulmonary tumor lesions.
  * In case of palliative irradiation to bone lesions in lung: at least 12 weeks must have passed at the date of registration since the last irradiation of the sites.
  * In case of irradiation to non-pulmonary sites: at least two weeks must have passed at the date of inclusion since the last irradiation of the sites
* At the time of registration, at least the following period has passed since last date of the prior therapy or procedure:

  * Surgery(including exploratory/ examination thoracotomy): 4 weeks
  * Pleural cavity drainage: 1 weeks
  * Pleurodesis without anti-neoplastic agents (inclusive of BRM such as Picibanil): 2 week
  * Biopsy accompanied by incision (including thoracoscopic biopsy): 2 week
  * Procedure for trauma (exclusive of patients with unhealed wound): 2 weeks
  * Transfusion of blood, preparation of hematopoietic factor: 2 week
  * Puncture and aspiration cytology: 1 week
  * Other investigational product: 4 weeks
* Written informed consent form

Exclusion Criteria:

* Previous history of malignancy within 3 years from study entry except treated non-melanomatous skin cancer, uterine cervical cancer in situ, or thyroid cancer
* Prior chemotherapy or systemic anti-cancer therapy for metastatic disease but postoperative adjuvant or neoadjuvant therapy of 6 months or more previously is allowed
* Patients who received previous treatment for lung cancer with drugs
* Symptomatic or uncontrolled central nervous system (CNS) metastases
* Patients with increased risk of bleeding, clinically significant cardiovascular diseases, a history of thrombosis or thromboembolism in the 6 months prior to treatment, gastrointestinal problems, and neurologic problems
* Any significant ophthalmologic abnormality
* Pre-existing parenchymal lung disease such as pulmonary fibrosis
* Known allergic history of Erlotinib or Bevacizumab
* Interstitial lung disease or fibrosis on chest radiogram
* Active infection, uncontrolled systemic disease (cardiopulmonary insufficiency, fatal arrhythmias, hepatitis)
* Pregnant or nursing women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to at least 36 months.
  Progression Free Survival

SECONDARY OUTCOMES:
ORR | through study completion, and average of 2 years
  Overall Response Rate
OS | From date of randomization until the date of death or date of last visit/contact, whichever came first, assessed to at least 36 months
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Youn Han, Ph.D, Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deng Z, Qin Y, Liu Y, Zhang Y, Lu Y. Role of Antiangiogenic Agents Combined With EGFR Tyrosine Kinase Inhibitors in Treatment-naive Lung Cancer: A Meta-Analysis. Clin Lung Cancer. 2021 Jan;22(1):e70-e83. doi: 10.1016/j.cllc.2020.08.005. Epub 2020 Sep 18. PMID 33067126